CLINICAL TRIAL: NCT07384299
Title: Impact of Baumann Skin Type on Wound Healing and Scar Formation Following Facial Skin Surgery
Brief Title: Impact of Skin Type on Wonud Healing and Scarring Following Facial Skin Surgery
Status: Completed | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, YangLiu82, Deputy Head of the Dermatology Department, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: WuhanUH-2025PFKBaumann
Record Dates: First submitted 2026-01-18; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Nevus; Seborrheic Keratosis (SK); Cyst; Lipoma; Scar
MeSH Terms: conditions — Nevus; Keratosis, Seborrheic; Cysts; Lipoma; Cicatrix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Oily Skin: classified as having oily skin according to the Baumann questionnaire
- Dry Skin: classified as having dry skin according to the Baumann questionnaire

SUMMARY:
The goal of this observational study is to learn how an individual's skin type influences the wound healing process and scar formation in Chinese patients undergoing facial dermatologic surgery. The main questions it aims to answer are:

How does skin type affect the quality of wound healing after facial surgery?

How does skin type affect the formation of hypertrophic scars after facial surgery?

Researchers will compare groups of patients with different skin types (classified by the Baumann Skin Type) to see if there are significant differences in their healing outcomes and scar characteristics.

Participants in this study will:

Receive standard facial dermatologic surgery as part of their clinical care.

Have their skin type assessed preoperatively.

Undergo scheduled postoperative follow-up assessments at 7 and 90 days to evaluate wound healing and scar development using standardized scales.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 14 and 60 years.
* Clinically and postoperatively pathologically diagnosed with a facial benign tumor (e.g., melanocytic nevus, sebaceous cyst, seborrheic keratosis, etc.) and having undergone standard surgical treatment.
* Voluntary participation in this study with written informed consent obtained.
* Commitment to comply with all study protocols and to complete all follow-up visits and data collection procedures.

Exclusion Criteria:

* Clinically or postoperatively diagnosed with a facial malignant tumor.
* Wounds requiring staged excision or planned for secondary intention healing.
* Surgical site located on or adjacent to the mucosal surface.
* Known history of allergy to any medications or dressings to be used during or after surgery.
* Presence of systemic diseases that significantly impair wound healing (e.g., poorly controlled diabetes, immunodeficiency disorders, active infections).
* Current use of medications affecting wound healing or scar formation (e.g., long-term systemic corticosteroids, immunosuppressants).
* Pregnancy or lactation.
* Refusal to provide written informed consent, or anticipated inability to comply with study follow-up and data collection.
* Concurrent participation in another interventional clinical trial.
* Any other condition deemed by the investigator as likely to interfere with study results or increase participant risk.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients undergoing facial skin surgery to remove benign lesions
Sampling Method: Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Patient and Observer Scar Assessment Scale version 2.0 (POSAS 2.0) | 3-month follow-up
  This scale comprises two separate subscales: the Observer Scar Assessment Scale (completed by the clinician) and the Patient Scar Assessment Scale (completed by the participant). The Observer Scale evaluates six items (vascularity, pigmentation, thickness, relief, pliability, and surface area) on a scale from 1 ("like normal skin") to 10 ("the worst scar imaginable"), with a total score ranging from 6 (best) to 60 (worst). The Patient Scale evaluates six items (pain, itching, color, stiffness, thickness, and irregularity) on a scale from 1 ("no, not at all") to 10 ("yes, very much"), with a total score also ranging from 6 (best) to 60 (worst). For both subscales, a higher score indicates a worse scar quality.
modified Stony Brook Scar Evaluation Scale (mSBSES) | 3-month follow-up
  Evaluations were independently performed by two clinicians who were blinded to group allocation. The scale comprises four items: scar width, height, color, and suture marks. Each item is scored from 0 to 2 points, where a score of 2 represents the closest resemblance to normal skin, and 0 represents the worst appearance. The total score ranges from 0 to 8, with a higher score indicating a more ideal scar appearance.

SECONDARY OUTCOMES:
Incidence of Postoperative Edema | 7-day follow-up
  Assessed by direct clinical examination. Unit: % of participants with the presence of edema.
Incidence of Wound Suppuration | Assessed by direct clinical examination. Unit: % of participants with the presence of suppuration.
  7-day follow-up
Incidence of Peri-wound Erythema | 7-day follow-up
  Assessed by direct clinical examination. Unit: % of participants with the presence of erythema.
Incidence of Wound Tenderness | 7-day follow-up
  Assessed by patient report. Unit: % of participants reporting tenderness.
Incidence of Postoperative Hemorrhage | 7-day follow-up
  Assessed by direct clinical examination. Unit: % of participants with active bleeding or hematoma formation.
Incidence of Peri-wound Ecchymosis | 7-day follow-uo
  Assessed by direct clinical examination. Unit: % of participants with the presence of ecchymosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Not Appicable, Wuhan, Hubei, China